CLINICAL TRIAL: NCT03270189
Title: Effect of the Visual Information Change in Functional Dystonia
Acronym: PRISMADYS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSA_2016_23
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Dystonia; Dystonic Disorders; Torticollis; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Dyskinesias; Neurologic Manifestations
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Torticollis; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Dyskinesias; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orthoptic treatment (Experimental): Patients with cervical dystonia occuring only during handwriting.
  Interventions: Device: prism glasses
- Controls (No Intervention): Patients without cervical dystonia.

INTERVENTIONS:
Device: prism glasses — orthoptic treatment by wearing prisms when writing
  Arms: orthoptic treatment

SUMMARY:
Cervical dystonia occurring only during the writing task is a rare form for which there is no established treatment. Many authors agree that alteration of sensory integration is associated with dystonia. Similar disturbances in the integration of oculomotor information could have a role in cervical dystonia forms involving visuo-cervico-manual coordination such as handwriting. We hypothesize that orthoptic treatment by wearing prisms when writing (i) will reduce the abnormal posture of the head occurring whilst writing and remove the associated nuchal pain; (ii) the correction after a period of systematic wearing of the prisms during handwriting tasks will have a sustainable effect allowing to keep a normal head position after the suppression of the prisms.

ELIGIBILITY:
Inclusion Criteria:

Case

* Presenting a cervical dystonia that occurs only during handwriting tasks, diagnosed by a neurologist specialised in movement disorders
* Being treated or not by injection of Botulinum Neurotoxin (but last injection > 3 months before the initial assessment)

Control

* No cervical dystonia
* Same sex, age (± 5 years), socio-professional level and hand laterality as the cases

Exclusion Criteria:

Case

* Cervical dystonia occuring in other circumstances than handwriting
* Neurological disease other than cervical dystonia (e.g. Parkinson's syndrome)
* Pain, trauma or pathology of the cervical spine of another cause than cervical dystonia and which have required medical or surgical treatment in the last 6 months preceding the initial assessment

Control

* Cervical disorders requiring medical or surgical treatment in the last 6 months prior to the tests
* Neurological disease affecting the cervical region or the writing hand
* Uncorrected visual disorders

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
measure of head movement occurring when writing | 3 months
  Difference of the angle measured with and without corrective prisms during the handwriting tasks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Bleton, PhD, Study Chair — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France